CLINICAL TRIAL: NCT06183814
Title: An Open-label, Dose-escalation Phase I/IIa Study to Evaluate the Safety and Efficacy of EXG102-031 Intraocular Injection in Participants With Neovascular Age-related Macular Degeneration（wAMD）
Brief Title: A Study of EXG102-031 in Participants With wAMD
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hangzhou Jiayin Biotech Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: EXG102-031-111
Record Dates: First submitted 2023-12-04; First posted 2023-12-28 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2024-01

CONDITIONS: Neovascular Age-related Macular Degeneration
Keywords: Wet Age-related Macular Degeneration

STUDY DESIGN:
Intervention Model Description: Dose escalation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Dose escalation-Cohort 1 (Experimental): Genetic : EXG102-031
  Interventions: Biological: EXG102-031
- Dose escalation-Cohort 2 (Experimental): Genetic : EXG102-031
  Interventions: Biological: EXG102-031
- Dose escalation-Cohort 3 (Experimental): Genetic : EXG102-031
  Interventions: Biological: EXG102-031
- Dose escalation-Cohort 4 (Experimental): Genetic : EXG102-031
  Interventions: Biological: EXG102-031
- Dose escalation-Cohort 5 (Experimental): Genetic : EXG102-031
  Interventions: Biological: EXG102-031

INTERVENTIONS:
Biological: EXG102-031 — EXG102-031 is a recombinant adeno-associated virus (rAAV) expressing an angiopoietin domain and VEGF receptor (ABD-VEGFR) fusion protein. EXG102-031 will be administered by subretinal injection.

SUMMARY:
In neovascular (wet) age-related macular degeneration (wAMD), the macula, or the part of the eye that provides the clear, detailed central vision, is being affected by abnormal blood vessel growth and leakage. This leakage affects the vision over time and can lead to severe blurriness or blinding. EXG102-031 was made to block the extra vessel formation which would lead to less leakage affecting the vision. Before EXG102-031 can be tested for its efficacy (if it makes vision better), it must be tested to see if it is safely tolerated to confirm it can continue to be studied in more patients with wAMD.

DETAILED DESCRIPTION:
Age-related macular degeneration (AMD) is a major cause of blindness and visual impairment in older adults. The wet form of AMD, also called neovascular AMD (nAMD) usually causes faster vision loss than the dry form. The most common current treatments of nAMD are products that inhibit vascular endothelial growth factor (VEGF) (including ranibizumab (LUCENTIS®, Genentech) and aflibercept (EYLEA®, Regeneron) and are delivered by intravitreal injections at 4 to 16 week intervals and continued indefinitely. This Open-label, Dose-escalation Phase I/IIa Study is designed to evaluate the safety and efficacy of EXG102-031 intraocular Injection in participants with wet(Neovascular) Age-related Macular Degeneration（wAMD）.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, age ≥ 50 years of age;
2. Diagnosis of wAMD and current active lesion in the study eye at Screening;
3. An ETDRS BCVA letter scores between 73 and 9 letters in the study eye;
4. Response to anti-VEGF treatment within 6 months prior to screening or at the time of screening introduction;
5. The study eye must be a Intraocular lens eye(post-cataract surgery status) and be at least 1 month post IOL implantation at enrollment;
6. Voluntarily agree to participate in the clinical trial, understand the trial procedures, and be capable of signing the informed consent form before screening.

Exclusion Criteria:

1. Presence of any ocular disease or history of disease in the study eye other than wAMD that may affect central visual acuity and/or macular detection;
2. Presence in the study eye of CNV or macular pathology pathography due to causes other than wAMD;
3. The study eye has severe and irreversible retinal structural damage involving the fovea (such as retinal pigment epithelial (RPE) atrophy, retinal fibrosis, laser scars, dense hard exudation); Or other retinal damage in the target eye that, in the opinion of the investigator, may impede visual improvement after resolution of macular edema ;
4. Subretinal hemorrhage accumulating the central fovea of the study eye, with an area of hemorrhage ≥ 4 optic disc diameters;
5. Presence of advanced glaucoma or uncontrolled ocular hypertension in the study eye;
6. Prior receipt of any ocular or systemic gene therapy agent.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2023-10-12 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety (Participants With Ocular and Non-ocular AEs (Adverse Events) and SAEs (Serious Adverse Events) | 24 weeks following EXG102-031 administration
  incidence of ocular and non-ocular AEs and SAEs

SECONDARY OUTCOMES:
Safety (Participants With Ocular and Non-ocular AEs (Adverse Events) and SAEs (Serious Adverse Events) | 52 weeks following EXG102-031 administration
  incidence of ocular and non-ocular AEs and SAEs
Change From Baseline in BCVA (Best Corrected Visual Acuity) | 52 weeks following EXG102-031 administration
  Visual function of the study eye was assessed using the Early Treatment Diabetic Retinopathy Study (ETDRS) Best Corrected Visual Acuity (BCVA) letter score. A higher score represents better vision.
Change From Baseline in CRT (Central Retinal Thickness) | 52 weeks following EXG102-031 administration
  Retinal fluid status of the study eye was evaluated using spectral domain OCT (Optical Coherence Tomography). A decrease in value indicates a decrease in fluid
Supplemental Injections (Annualized Rate of Supplemental Injections) | 52 weeks following EXG102-031 administration
  The number of supplemental anti-VEGF injections given after EXG102-031 was administered.

CONTACTS AND LOCATIONS:
Overall Officials: Mingwei Zhao, PhD, Principal Investigator — Peking University People's Hospital
Locations (8):
- China (8):
  - Beijing Hospital, Beijing, Beijing Municipality
  - Beijing Tongren Hospital,Cmu, Beijing, Beijing Municipality
  - Peking University People'S Hospital, Beijing, Beijing Municipality
  - The Southwest Hospital of Amu, Chongqing, Chongqing Municipality
  - Central theater General Hospital, Wuhai, Hubei
  - Jiangsu Provinve Hospital, Nanjing, Jiangsu
  - The Second Affiliated Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Eye Hospital,WMU, Wenzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No